CLINICAL TRIAL: NCT05882968
Title: Prevalence of Helicobacter Pylori in Chronic Kidney Diseases in Assiut University Hospitals
Brief Title: Prevalence of H.Pylori in CKD Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, hanaa zakaria william, resident of nephrology, Assiut University
Other Study IDs: H.pylori in CKD patients
Record Dates: First submitted 2023-05-14; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: H.Pylori Infection
Keywords: CKd patients
MeSH Terms: interventions — Kidney Function Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- H. Pylori in CKD patients: 100 0f patients with H.pylori with ckd according to GFR more than 60 according to kdigo guide lines
  Interventions: Diagnostic Test: kidney function tests
- H.pylori in normal renal function: 100 of patients with H.pylori with normal renal function according to GFR less than 60 according to kdigo guide lines

INTERVENTIONS:
Diagnostic Test: kidney function tests — using GFR test according to kdigo guide lines
  Groups: H. Pylori in CKD patients

SUMMARY:
The study aims to:-

- Investigate the relationship between H. pylori and CKD, in order to determine whether an association exists between H.pylori and kidneys.

DETAILED DESCRIPTION:
Helicobacter pylori is a spiral-shaped, gram-negative flagellated bacterium that usually resides in the gastric mucosa [1]. It affects approximately 50% of the world's population, even 80% in lower and middle outcome countries [1] [2].

The prevalence according to a study conducted by Ankouane et al. in Yaoundé (Cameroon) is up to 72.5% in hospital [3]. The main route of transmission is person to person transmission and often occurs in the first 5 years of life [4].

Helicobacter pylori is the most common human chronic infection, causing gastrointestinal diseases such as gastric malignancies, gastritis, and ulcerative diseases. H. pylori can also be involved in other non-gastrointestinal infections such as diabetes and metabolic syndrome, heart disease, hematologic disorders, cancer, and chronic kidney disease (CKD) as well as chronic renal failure (CRF) [5].

The risk factors for infection with H. pylori are low socioeconomic level, promiscuity, family history of H. pylori infection or gastritis, alcohol consumption, smoking [6].

The stomach is reported to be associated with conditions affecting other organs. Such as, an association between atrophic gastritis (AG) and coronary artery disease has been described, with AG representing a potential independent risk factor for coronary artery disease [7].

The diagnosis of H. pylori is made by noninvasive methods (the rapid urease test, the breath test, serology, stool antigen test) or invasive methods biopsy-based tests (culture and histology) [8]. The gold standard is histology, but current methods have been developed, using high-definition endoscopy [9].

Chronic kidney disease (CKD) is a growing disease and public health problem worldwide [10]. Gastrointestinal (GI) symptoms are common among subjects with CKD, and their intensity vary slightly to very severe, altering the quality of life and potentially hindering the effectiveness of the treatment [11] and also affects their nutrition status leading to the development of malnutrition, which is a potent predictor of morbidity and mortality [12].

Patients with chronic renal failure (CRF) often have gastrointestinal symptoms caused not only by H. pylori infection, but also by high urea levels, decline of gastrointestinal motility, hypergastrinemia and high ammonia levels [10-13].

Moreover, patients with CRF may have higher risks of gastric mucosal damages compared with individuals with normal renal function because of systemic and/or local chronic circulatory failure [14].

Epidemiological studies have revealed a link between H. pylori with insulin resistance and metabolic syndrome , which may increase the risk of CKD. However, up to date there is no conclusive evidence regarding the association between H. pylori infection and CKD [15].

A previous study reported that individuals infected with H. pylori had a higher risk of subsequent renal dysfunction than those not infected [12]. Conversely, the H. pylori infection rate is lower in patients with peptic ulcer disease and concomitant chronic kidney disease (CKD) than in those without CKD [13]. However, the relationship between H. pylori infection and/or gastric disorders and CKD has not been elucidated.

ELIGIBILITY:
Inclusion Criteria:

* Patients age >18 -65 years.

  * 100 of them are CKd with GFR less than 60 according to kdigo guidelines
  * 100 of them are normal renal function with GFR more than 60 according to kdigo guidelines

Exclusion Criteria:

* • H-pylori eradication

  * History of gastrectomy
  * Used proton-pump inhibitor. Patients with Past or present history of malignancy

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 200 of patients with H. pylori
  100 of them with ckd
  100 of them with normal renal function
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Relationship between H.pylori and CKD patients according to Glomural filtration rate (GFR )according to kdigo guide lines | july 2023 to july 2025
  To assess if H pylori with CKd patients more than H pylori in normal renal function patients or not that aging 18_65 years

CONTACTS AND LOCATIONS:
Overall Officials: Abd elhamid Mohammed, Study Director — Assiut University